CLINICAL TRIAL: NCT06684379
Title: Double-blind, Randomized, Placebo-controlled, Pilot Clinical Trial to Evaluate the Safety, Tolerability and Efficacy of Two Doses of a Conditioned Medium From a Co-culture of M2-macrophages and Fat-derived Mesenchymal Cells (PRS CK STORM) in the Modulation of the Cytokine Storm for the Treatment of Acute Respiratory Distress Syndrome (ARDS) Caused by SARS-Cov-2, Influenza A, Influenza B and Respiratory Syncytial Virus (RSV)
Brief Title: Study on Safety and Efficacy of Two Doses of PRS CK STORM in the Modulation of the Cytokine Storm for the Treatment of Acute Respiratory Distress Syndrome (ARDS) Caused by SARS-Cov-2, Influenza A, Influenza B and Respiratory Syncytial Virus (RSV)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PEACHES BIOTECH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: PRSCK-21P01; 2023-507700-32-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-23; First posted 2024-11-12 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: SARS-CoV-2; Influenza, Human; Respiratory Syncytial Virus Infections; Respiratory Distress Syndrome
Keywords: SARS-CoV-2 infection; Causing atypical respiratory disease (COVID-19); 2019 Novel Coronavirus; COVID-19 Virus; SARS Coronavirus 2; COVID-19-associated cytokine storm; Lung Diseases; Pneumonia; M2-macrophages; Mesenchymal cells; Influenza A Virus; Influenza B Virus; RSV Infection; Acute Respiratory Distress Syndrome; ARDS, Human; Respiratory Distress Syndrome, Acute; Cytokine storm
MeSH Terms: conditions — Influenza, Human; Respiratory Syncytial Virus Infections; Respiratory Distress Syndrome; COVID-19; Lung Diseases; Pneumonia; Cytokine Release Syndrome | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in blocks; the study will be conducted in 2 parts in sequential groups of two increasing doses of PRS CK STORM (A and B) and consecutively evaluated in 2 sentinel groups of 4 patients. Patients will be randomized to receive treatment in groups of 2, for 5 consecutive days, until 48 hours after the last drug administration (short-term safety follow-up period).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Saline Solution 0,9% for injection (Active Comparator): Participants will receive a single 10 mL dose Intravenous (IV) infusion of normal saline (0.9%)
  Interventions: Drug: Placebo comparator
- PRS CK STORM - dose A (Experimental): A sterile secretome derived from the co-culture of M2-type macrophages and ASC (adipose stromal cells) containing 116,059 pg/mL Tissue Inhibitor of Matrix Metalloproteinase- 1 (TIMP-1). Participants will receive a total dose of 1,160,585.366 pg of TIMP-1 via IV infusion
  Interventions: Drug: PRS CK STORM
- PRS CK STORM - dose B (Experimental): A sterile secretome derived from the co-culture of M2-type macrophages and ASC (adipose stromal cells) containing 232,017 pg/mL TIMP-1. Participants will receive a total dose of 1,160,585.366 pg of TIMP-1 via IV infusion.
  Interventions: Drug: PRS CK STORM

INTERVENTIONS:
Drug: Placebo comparator — A single dose of saline solution 0.9% for infusion
  Other Names: Saline Solution
  Arms: Saline Solution 0,9% for injection
Drug: PRS CK STORM — A single dose of PRS CK STORM (dose A) for infusion
  Arms: PRS CK STORM - dose A
Drug: PRS CK STORM — A single dose of PRS CK STORM (dose B) for infusion.
  Arms: PRS CK STORM - dose B

SUMMARY:
The purpose of this clinical trial is to evaluate the safety, tolerability and efficacy of two doses (dose A and dose B) of Standardized Conditioned Medium Obtained by Coculture of Monocytes and fat-derived Mesenchymal Stromal Cells (PRS CK STORM) in the modulation of the cytokine storm for the treatment of the acute respiratory distress syndrome (ARDS) caused by SARS-Cov-2, influenza A, influenza B and respiratory syncytial virus (RSV) in recently hospitalized participants (less than 3 days) in need for oxygen therapy.

The main questions it aims to answer are:

* Are both doses of PRS CK STORM (dose A and dose B) safe as an intravenous drug to modulate inflammatory processes, such as the cytokine storm for the treatment of ARDS caused by SARS-Cov-2, influenza A, influenza B and RSV?
* Are both doses of PRS CK STORM (dose A and dose B) effective as an intravenous drug to modulate ARDS-associated cytokine storm caused by SARS-Cov-2, influenza A, influenza B and RSV compared to the control group?
* What are the anti-inflammatory and pro-inflammatory cytokine profiles after treatment with two different doses of PRS CK STORM in participants hospitalized for ARDS caused by SARS-Cov-2, influenza A, influenza B and RSV?

Researchers will compare both doses of PRS CK STORM with the control group to test whether the anti-inflammatory action of PRS CK STORM is safe and effective in modulating the cytokine storm for the treatment of ARDS caused by SARS-Cov-2, influenza A, influenza B and RSV. In addition, the anti-inflammatory and pro-inflammatory cytokine profiles after treatment PRS CK STORM compared to placebo group in these participants will be also studied.

DETAILED DESCRIPTION:
This is a double-blind, randomized, phase I/II pilot clinical trial of two doses of PRS CK STORM in hospitalized adult participants with ARDS caused by SARS-Cov-2, influenza A, influenza B and RSV All participants will receive the standard of care for ARDS, according to its viral origin:

* Clinical management of COVID-19: hospital care (Centro de Coordinación de Alertas y Emergencias Sanitarias, 2020).
* Clinical practice guidelines for influenza (WHO, 2024). Participants who meet the eligibility criteria will be randomized in blocks to reach the 2:2:1 ratio (dose A: dose B: placebo).

This study consists of two parts:

Part 1: Two different doses (A and B) of PRS CK STORM will be evaluated in 2 groups of 4 participants (3:1; PRS CK STORM: placebo). It starts with a first sentinel group of 4 participants who will be assigned to placebo or study drug dose A. First, only 2 participants will randomly be assigned to receive the active treatment of dose A or placebo for 5 consecutive days. These 2 first participants will be followed up to 48h after the last drug administration (short-term safety follow-up period) when a safety assessment will be completed before treating the other 2 participants in this group.

If the study drug is considered safe during the short-term safety assessment planned 48h after the last drug administration, then 2 additional participants will be treated with dose A for 5 consecutive days to complete the first sentinel group of 4 participants. These 2 participants will be followed up to 48h after the last study drug administration before moving to dose B.

After the assessment of data collected follow-up for this first group, a second small sentinel group of other 4 participants will be treated with a higher dosage (dose B) following the same process: firstly, only 2 participants will randomly receive the active treatment of dose B or placebo for 5 consecutive days and then these 2 first participants will be followed up to 48h after.

If the study drug is considered safe during the safety assessment planned 48h after last drug administration, then two additional participants will be treated with dose B for 5 consecutive days to complete the sentinel second group of 4 participants evaluating dose B. These 2 participants will be also followed up to 48h after the last study drug administration before moving to Part 2.

All these 8 participants included in Part 1 will continue in a long-term safety follow-up period until 1 year post treatment.

Part 2: 42 additional participants will be treated for 5 consecutive days. These 42 participants will be randomized to three treatment arms: 17 in the active arm with dose A, 17 participants in the active arm with dose B and 8 participants in the placebo arm. All participants in Part 2 will be followed up to 48h after the last study drug (short-term safety follow-up period). Once all participants treated in Part 2 finished the short-term safety follow-up period (48h after last study drug administration), all data will be verified and statistically analyzed in an interim analysis. All participants will be followed up to 1 year post treatment (long-term safety follow-up period). Therefore, considering the participants enrolled in Part 1 and Part 2 the total number of participants for safety, tolerability and efficacy analysis will be 50 assigned to three different arms (total randomization ratio 2:2:1), 20 participants will receive dose A, 20 participants will receive dose B and 10 participants will receive placebo.

To sum up, considering the participants enrolled in Part 1 and Part 2 the total number of participants for safety, tolerability and efficacy analysis will be 50 assigned to three different arms (total randomization ratio 2:2:1), 20 participants will receive dose A of PRS CK STORM, 20 participants will receive dose B of PRS CK STORM and 10 participants will receive placebo.

The estimated duration of the study for individual participants will be 12 months (screening: 3 days, treatment period: 5 days, short-term safety follow-up period: 2 days after the last drug intake and long-term safety follow-up period: up to 48 weeks from randomization).

It is hypothesized that both doses of PRS CK STORM for intravenous administration are safe, well tolerated and clinically beneficial versus placebo for participants with ARDS-associated cytokine storm.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent by the patient or legal representative prior to the initiation of any study-specific procedure.
2. Males and females aged ≥ 18 years old at the time of the consent.
3. Hospitalized patients with a diagnosis of ARDS confirmed by Berlin criteria.
4. Confirmed diagnosis of SARS-CoV-2, influenza virus A, influenza virus B or RSV pneumonia by positive RT-PCR (results of a PCR prior to screening will be valid only if the PCR has been done for all 4 viruses and in 3 days prior to the screening visit). PCR will include the analysis of SARS-Cov-2, influenza A, influenza B and RSV.
5. Diagnosis of systemic inflammatory response syndrome (SIRS), defined by the satisfaction of any two of the criteria below:

   1. Body temperature over 38 ºC or under 36 ºC.
   2. Heart rate greater than 90 beats/minute.
   3. Respiratory rate higher than 20 breaths/min or PaCO2 lower than 32 mmHg.
   4. Leukocyte count higher than 12000/μL, lower than 4000/μL or over 10% immature forms or bands.
6. Need for oxygen therapy.
7. Participants to be hospitalized or who have been admitted for less than 3 days and who have had symptoms up to a maximum of 10 days prior to screening.
8. Female participants must be, either surgically sterilized or at least 1 year postmenopausal (confirmed by follicle-stimulating hormone [FSH] more than 20 international units [Ius] only for women under 54) or using adequate birth control (hormonal contraception, intrauterine contraceptive device, double barrier methods [condom with spermicide, diaphragm with spermicide, or condom and diaphragm]) or sexual abstinence for up to 90 days after the last treatment administration. Male participants must be willing to use barrier contraception (condom) for up to 90 days after the last treatment administration.

Exclusion Criteria:

1. Failure to perform screening or baseline examinations.
2. Body Mass Index (BMI) more than or equal to 35.
3. Irreversible critical condition.
4. Active autoimmune diseases or severe immunosuppression.
5. Clinically significant, advanced or unstable disease that may interfere with primary or secondary variable evaluations, may bias the clinical assessment, such as:

   1. Liver function test abnormalities or other signs of hepatic insufficiency: Aspartate transaminase (AST), alanine transaminase (ALT) more than 3 per upper limit of the reference range, total bilirubin more than or equal to 2 mg/dL; except for subjects with isolated elevation of indirect bilirubin relating to Gilbert syndrome.
   2. Renal insufficiency (serum creatinine more than 2 mg/dL (more than 150 μmol/L) and creatinine clearance less than 60 (according to Cockcroft-Gault formula).
   3. Myocardial infarction, unstable angina, heart failure within 3 months before screening.
   4. Bradycardia (heartbeat less than 50/min).
   5. Atrioventricular block (type II / Mobitz II and type III), congenital long QT syndrome, sinus node dysfunction or prolonged QTcF interval (males more than 450 msec and females more than 470 msec using Fridericia's formula: QTc = QT/ RR^2 ).
   6. Uncontrolled diabetes mellitus (blood glucose level above 500 mg/dL) at the time of admission.
   7. Malignant tumors within the last 5 years except skin malignancies (other than melanoma) or indolent prostate cancer
   8. Metastases.
   9. Human Immunodeficiency Virus (HIV), HBV [hepatitis B surface antigen (HBs Ag) positive (+), or detected sensitivity on the HBV deoxyribonucleic acid (DNA), polymerase chain reaction (PCR) qualitative test for hepatitis B core antibody (HBc Ab) positive subjects] or HCV [HCV ribonucleic acid (RNA) detectable in any subject with positive anti-HCV antibody (HCV Ab)].
   10. Other serious active viral infections apart from SARS-CoV-2, influenza A, influenza B or RSV that require specific antimicrobial treatment.
6. Inability to comply with the study and monitoring procedures.
7. Pregnant and breastfeeding females (pregnancy test positive).
8. Suspected or known history of drug or alcohol abuse.
9. Enrollment in another investigational drug study within 1 month before the screening
10. Subject who has any condition, including any psychological or psychiatric condition, in the opinion of the Investigator, would compromise the safety of the subject or the quality of the data and renders the subject an unsuitable candidate for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2026-10-02 (Estimated); Study Completion 2026-10-02 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AEs) | Up to 12 months
  Number and proportion of subjects experiencing AEs.
Serious adverse events (SAEs) | Up to 12 months
  Number and proportion of subjects experiencing SAEs
Treatment-emergent adverse events (TEAEs) | Up to 12 months
  Number and proportion of subjects experiencing TEAEs
Safety measures: Clinical evaluation through physical examination | Day 7, Day 30, Day 90 and Day 365
  Number and proportion of subjects with abnormal findings of physical examination parameters (head, ears, Nervous system,Gastrointestinal system, Respiratory system, Lymph nodes Musculoskeletal system, Neck, Throat, Cardiovascular system, Skin, Nose) will be evaluated
Changes from Baseline in vital signs: body temperature | From Day 1 to Day 7, Day 30, Day 90 and Day 365
  Body Temperature of participants will be measure d in Celsius (ºC)
Changes from Baseline in vital signs: oximetry | From Day 1 to Day 7, Day 30, Day 90 and Day 365
  Levels of blood oxygen saturation (SpO2) using a pulse oximeter will be measured in percentage
Changes from Baseline in vital signs: Heart rate | From Day 1 to Day 7, Day 30, Day 90 and Day 365
  Heart rate will be measured as number of beats per minute (bpm)
Changes from Baseline in vital signs: Respiratory rate | From Day 1 to Day 7, Day 30, Day 90 and Day 365
  Respiratory rate will be measured as number of breaths taken per minute (Breaths/min) .
Changes from Baseline in vital signs: Diastolic Blood Pressure | From Day 1 to Day 7, Day 30, Day 90 and Day 365
  Diastolic blood pressure will be measured in mmHg
Changes from Baseline in vital signs: Systolic blood pressure | : From Day 1 to Day 7, Day 30, Day 90 and Day 365
  Systolic blood pressure will be measured in mmHg
Safety measures: electrocardiograms (ECG) | Day 7, Day 30, Day 90 and Day 365
  Cardiac dysfunction will be monitored by 12-lead ECGs. Abnormal or normal readings will be evaluated
Safety measures: Laboratory results | Day 1, Day 3, Day 6, Day 7, Day 30, Day 90 and Day 365
  Abnormal or normal laboratory test results (biochemistry, hematology, coagulation, and urinalysis) will be evaluated

SECONDARY OUTCOMES:
Severity of ARDS | Up to 12 months
  Severity of ARDS will be assessed as the values of the Kirby index (ratio PaO2/FiO2). Severity according to PaO2/FiO2 values is classified as:
  * Normal: PaO2/FiO2 > 300 mmHg
  * Mild: 200 mmHg < PaO2/FiO2 ≤ 300 mmHg
  * Moderate: 100 mmHg < PaO2/FiO2 ≤ 200 mmHg
  * Severe: PaO2/FiO2 ≤ 100 mmHg
Death rate | Day 7, Day 14 and Day 365
  Percentage of participants who died since the beginning of treatment. Death rate at each timepoint will be studied by means of a difference between independent proportions tests
Average hospital stays (in days) | Up to 12 months
  Average of days that participants stay in the hospital
Participants requiring admission to Intensive Care Unit (ICU) | Up to 12 months
  Percentage of participants requiring admission to ICU
Duration of ICU stay | Up to 12 months
  Average of days that participants stay in ICU
Thorax radiological findings | Day 7 and Day 10 Up to 12 months
  Percentage of participants with the following thorax radiological findings:
  * Pneumonia (unilateral, bilateral).
  * Infiltrates.
  * Stabilization.
  * radiological evolution.
Oximetry levels | Up to 12 months
  Changes in the levels of blood oxygen saturation.
Overall survival (in days) | Up to 12 months
  Proportion of participants who survive the disease during the follow-up period
Time to progression (in days) | Up to 12 months
  Period from the initiation of treatment until the detection of disease progression or worsening symptoms in a patient with COVID-19.
Need for invasive mechanical ventilation | Up to 12 months
  The need of the use of a ventilation machine to fully or partially provide artificial ventilation via an invasive procedure such as intubation (endotracheal tube) or tracheostomy (tracheostomy tube) will be evaluated.
Time to invasive mechanical ventilation (in days) | Up to 12 months
  Period of time (in days) under need of the use of a ventilation machine to fully or partially provide artificial ventilation via an invasive procedure such as intubation (endotracheal tube) or tracheostomy (tracheostomy tube).

OTHER OUTCOMES:
Variations in anti-inflamatory cytokine levels | Day 1, Day 3 and Day 6
  Changes in the concentrations of anti-inflammatory (TIMP-1 and IL-1Ra) cytokines before and after treatment. Blood samples will be collected from patients to carry out cytokine quantification
Variation in pro-inflammatory cytokine levels | Day 1, Day 3 and Day 6
  Changes in the concentrations of pro-inflammatory (TNF-α, IL-1β, IL-6 and IL-18) cytokines before and after treatment. Blood samples will be collected from patients to carry out cytokine quantification.

CONTACTS AND LOCATIONS:
Overall Officials: David Bernal, Dr., Principal Investigator — Hospital Universitario de Fuenlabrada; Guillermo Soria Fernández-Llamazares, Dr, Study Chair — Hospital Universitario de Fuenlabrada
Locations (1):
- Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lapuente JP, Gomez G, Marco-Brualla J, Fernandez P, Desportes P, Sanz J, Garcia-Gil M, Bermejo F, San Martin JV, Algaba A, De Gregorio JC, Lapuente D, De Gregorio A, Lapuente B, Gomez S, Andres MLV, Anel A. Evaluation in a Cytokine Storm Model In Vivo of the Safety and Efficacy of Intravenous Administration of PRS CK STORM (Standardized Conditioned Medium Obtained by Coculture of Monocytes and Mesenchymal Stromal Cells). Biomedicines. 2022 May 8;10(5):1094. doi: 10.3390/biomedicines10051094. PMID 35625831
- [Background] Centro de Coordinación y Alertas Sanitarias (coord.). Manejo clínico del COVID-19: atención hospitalaria. Madrid: Ministerio de Sanidad; 2020.
- [Background] Clinical practice guidelines for influenza [Internet]. Geneva: World Health Organization; 2024. Available from http://www.ncbi.nlm.nih.gov/books/NBK607904/ PMID 39374347
- [Result] Lapuente JP, Blazquez-Martinez A, Marco-Brualla J, Gomez G, Desportes P, Sanz J, Fernandez P, Garcia-Gil M, Bermejo F, San Martin JV, Algaba A, De Gregorio JC, Lapuente D, De Gregorio A, Lapuente B, Andres MV, Anel A. Cytokine Profile and Anti-Inflammatory Activity of a Standardized Conditioned Medium Obtained by Coculture of Monocytes and Mesenchymal Stromal Cells (PRS CK STORM). Biomolecules. 2022 Mar 31;12(4):534. doi: 10.3390/biom12040534. PMID 35454123